CLINICAL TRIAL: NCT01439139
Title: Portable Bone Ultrasonometer for Osteoporosis Assessment
Brief Title: Bone UltraSonic Scanner (BUSS): Validation Study
Status: Completed | Type: Observational
Sponsor: Artann Laboratories (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: BUSS-04; 2R44AG017400 (NIH)
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Osteoporosis; Osteopenia
Keywords: Osteoporosis; ultrasound; sonometer; DXA
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of clinical study is to assess effectiveness of Bone UltraSonic Scanner (BUSS) versus densitometry (DXA) in osteoporosis detection.

DETAILED DESCRIPTION:
Study will conduct measurements in a group of postmenopausal women and use their DXA examination data as a control. BUSS data will be able to discriminate between postmenopausal women with osteoporosis compared with no osteoporosis defined by DXA measurements.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* Age 50-90 years
* Any race or ethnicity
* DXA spine and hip exam within one year

Exclusion Criteria:

* Open wounds or rashes on the testing area
* Active skin infection
* Recent tibia surgery
* Abnormal tibia anatomy
* Body Mass Index > 34.9 kg/m2
* Current or previous tibial fracture on side of testing
* Stroke or with total or partial paralysis with residual disability lasting more than 3 months

Current or recent (within past 6 months) use of bone-active drugs:

* Bisphosphonates
* Calcitonin
* Estrogens or selective estrogen receptor modulator (SERM)
* Therapeutic doses of fluoride (> 2mg/day)
* Teriparatide used currently or within past 3 months
* Drugs under research protocols, and
* Unstudied or unapproved drugs
* Presence of metabolic bone disease

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
BUSS data will be able to discriminate between postmenopausal women with osteoporosis compared with no osteoporosis defined by DXA measurements. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Armen Sarvazyan, Ph.D., D.Sc., Study Chair — Artann Laboratories, Inc
Locations (1):
- Catholic Health System Affiliates & Sister's of Charity Hospital, Buffalo, New York, United States